CLINICAL TRIAL: NCT07270770
Title: A Single-center, Open-label, Investigator-Initiated Trial to Evaluate the Safety, Pharmacokinetics, and Efficacy of Menin Inhibitor BY002 in Patients With Relapsed or Refractory Acute Leukemia
Brief Title: BY002 IIT Study in R/R Acute Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chen Suning, Doctor, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2nd_Menin inhibitor
Record Dates: First submitted 2025-10-02; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Acute Leukemia; KMT2A Rearrangements or NPM1 Mutations Acute Leukemia
Keywords: KMT2A rearrangements or NPM1 mutations; relapsed or refractory acute leukemia; Menin Inhibitor
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BY002 treatment (Experimental): BY002 capsule (oral)
  * Starting dose: 50 mg BID
  * Dose escalation: 100 mg BID → 150 mg BID → 200 mg BID (3+3 design)
  * Treatment cycle: 28 days, repeated until disease progression, unacceptable toxicity, HSCT, withdrawal, or death
  Interventions: Drug: BY002

INTERVENTIONS:
Drug: BY002 — BY002 capsule (oral)
  * Starting dose: 50 mg BID
  * Dose escalation: 100 mg BID → 150 mg BID → 200 mg BID (3+3 design)
  * Treatment cycle: 28 days, repeated until disease progression, unacceptable toxicity, HSCT, withdrawal, or death

SUMMARY:
This is a single-center, open-label, investigator-initiated phase 1 study designed to evaluate the safety, pharmacokinetics (PK), and preliminary efficacy of the menin inhibitor BY002 in patients with relapsed or refractory acute leukemia. Eligible subjects include adult patients (≥18 years) with AML, ALL, or MPAL, excluding APL, who carry KMT2A rearrangement or NPM1 mutation and have no better treatment options.

The study will be conducted in a dose-escalation design (3+3) with an accelerated titration at the starting dose, followed by expansion at the recommended dose. BY002 is administered orally in 28-day cycles until disease progression, unacceptable toxicity, HSCT, withdrawal, or death.

The primary objectives are to determine the incidence of dose-limiting toxicities (DLTs) and serious adverse events (SAEs), and to define the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D). Secondary objectives include characterization of PK parameters, evaluation of safety (AEs, laboratory tests, vital signs, ECG), and assessment of efficacy endpoints such as complete remission (CR), composite remission (CRc), overall response rate (ORR), duration of response (DOR), event-free survival (EFS), relapse-free survival (RFS), overall survival (OS), and cumulative incidence of relapse (CIR). Exploratory objectives include analysis of pharmacodynamic biomarkers (e.g., HOXA9, MEIS1, CD11b) and correlation of baseline genetic mutations (e.g., NPM1, KMT2A, FLT3, TP53, NUP98) with clinical outcomes.

DETAILED DESCRIPTION:
Relapsed/refractory (R/R) acute leukemia remains a severe disease with poor prognosis, and current treatment options are limited. Patients carrying genetic alterations such as KMT2A rearrangements or NPM1 mutations are particularly challenging, as these mutations are associated with high relapse rates and treatment resistance. Existing therapies have shown limited benefit in this population, highlighting an urgent unmet need for novel targeted approaches.

BY002 is a selective menin inhibitor developed in China. Preclinical studies have demonstrated that menin inhibition can downregulate leukemogenic genes such as HOXA9 and MEIS1, induce differentiation, and restore sensitivity to treatment. Importantly, BY002 shows potential to overcome resistance driven by existing mutations including KMT2A rearrangements and NPM1 mutations, thereby offering a new therapeutic strategy for these high-risk patients.

This study is a single-center, open-label, investigator-initiated phase 1 trial designed to evaluate the safety, pharmacokinetics (PK), and preliminary efficacy of BY002 in adult patients with relapsed or refractory acute leukemia. The trial adopts a 3+3 dose-escalation design with accelerated titration at the starting dose, followed by expansion at the recommended dose.

Patients will receive oral BY002 in 28-day cycles until disease progression, unacceptable toxicity, hematopoietic stem cell transplantation, withdrawal, or death. Safety assessments will include the incidence of dose-limiting toxicities (DLTs), serious adverse events (SAEs), and overall adverse events, as well as laboratory tests, vital signs, and ECG monitoring. PK will be assessed by plasma concentrations of BY002 and its metabolite M1, together with parameters such as Cmax, Tmax, t1/2, AUC, CL/F, and V/F.

Secondary endpoints will evaluate efficacy according to ELN 2022 criteria, including complete remission (CR), composite remission (CRc), overall response rate (ORR), duration of response (DOR), event-free survival (EFS), relapse-free survival (RFS), overall survival (OS), and cumulative incidence of relapse (CIR). Exploratory analyses will assess changes in pharmacodynamic biomarkers (e.g., HOXA9, MEIS1, CD11b) before and after treatment, and investigate the correlation between baseline genetic alterations (such as KMT2A rearrangement, NPM1 mutation, FLT3 mutation/fusion, TP53 mutation, or NUP98 fusion) and clinical outcomes.

This trial will generate first-in-human data on BY002 in relapsed/refractory acute leukemia and provide essential evidence to guide subsequent phase 2/3 clinical development.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Confirmed diagnosis of AML, ALL, or MPAL per WHO 2022 criteria.
* Relapsed or refractory disease after ≥1 prior therapy.
* Presence of KMT2A rearrangement or NPM1 mutation (preferred, but not exclusive).
* ECOG performance status 0-2.
* Adequate organ function:
* ANC ≥1.0 × 10⁹/L (unless cytopenia due to leukemia)
* Platelets ≥50 × 10⁹/L (unless due to leukemia)
* ALT/AST ≤2.5 × ULN, bilirubin ≤1.5 × ULN
* Creatinine clearance ≥50 mL/min
* Negative pregnancy test for women of childbearing potential.
* Willing to use effective contraception during study and 90 days after last dose.
* Signed informed consent.

Exclusion Criteria:

* Active central nervous system (CNS) leukemia. (Prior CNS involvement allowed if treated and controlled; CNS prophylaxis permitted.)
* History of significant liver disease, including viral hepatitis or cirrhosis:
* HBsAg positive must have negative HBV DNA.
* HCV antibody positive must have negative HCV RNA.
* Known HIV infection.
* Pregnant or breastfeeding women.
* Significant cardiac disease:
* Congenital long QT syndrome or QTcF >450 msec.
* Acute myocardial infarction, unstable angina, or coronary artery bypass within 6 months.
* Congestive heart failure ≥ NYHA class II.
* History of another malignancy within 5 years, except adequately treated basal cell carcinoma of the skin, in-situ breast cancer, or in-situ cervical cancer.
* Autologous HSCT or CAR-T therapy within 60 days, or unresolved toxicities from ASCT/CAR-T.
* Allogeneic HSCT within 100 days, or active GVHD, or requiring ongoing immunosuppressive therapy.
* Anti-leukemia therapy within 2 weeks before study entry (hydroxyurea permitted).
* Prior investigational drug use: <2 weeks or <5 half-lives for small molecules; <4 weeks or <5 half-lives for biologics (whichever is shorter).
* Unresolved toxicities > grade 1 from prior anti-leukemia therapy (except alopecia).
* Uncontrolled active infection:
* Mild infections manageable with oral/topical treatment are allowed.
* Serious infections requiring hospitalization/IV antibiotics within 14 days excluded, unless resolved.
* Febrile neutropenia without infection evidence may be eligible if afebrile >72 h without antipyretics.
* Active tuberculosis excluded.
* Conditions impairing oral intake or absorption (e.g., swallowing difficulty, short bowel syndrome, gastroparesis).
* Known severe allergy to Menin inhibitors or any component of BY002.
* Investigator judges poor compliance or inability to complete study.
* Any other serious disease, abnormality, or condition that may increase risk, interfere with study drug, confound results, or expected survival ≤6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLT) | From Cycle 1 Day 1 (C1D1) through the end of the DLT observation period (Day 1-28; may extend to Day 42 if toxicity evaluation is delayed).
  A DLT is defined as any ≥Grade 3 non-hematologic or ≥Grade 4 hematologic toxicity considered related to BY002, occurring during the DLT evaluation period. The number and proportion of participants with DLTs will be summarized.
Incidence of serious adverse events (SAEs) | From Cycle 1 Day 1 (C1D1) until 30 days after the last dose.
  SAEs will be defined and classified according to ICH E2A and CTCAE v5.0. The number and proportion of participants experiencing ≥1 SAE will be summarized.

SECONDARY OUTCOMES:
Incidence, type, and severity of all adverse events (AEs) | From first dose until 30 days after the last dose.
  AEs will be coded per MedDRA and graded by NCI CTCAE v5.0. Number, type, severity, and causality of AEs will be summarized.
Plasma concentrations of BY002 and its primary metabolite (M1) | Cycle 0 Day 1 (single-dose PK) and throughout treatment cycles, up to 30 days after the last dose.
  PK parameters including Cmax, Tmax, AUC, t1/2, and CL/F will be calculated using non-compartmental analysis following single-dose and multiple-dose administration.
Proportion of participants achieving complete remission (CR/CRi) per ELN 2022 criteria | From first dose until disease progression, relapse, or death, assessed up to approximately 24 months.
  Response will be evaluated according to ELN 2022 criteria, including CR, CRi, PR, and MRD negativity rates.

OTHER OUTCOMES:
Pharmacodynamic biomarker changes and correlation of baseline genomic mutations with clinical efficacy | From baseline until end of study (up to 24 months).
  Quantitative assessment of pharmacodynamic markers (e.g., HOXA9, MEIS1 expression) and exploratory analysis of association between baseline mutation profiles and treatment response or survival outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Suning Chen, MD, PhD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided